CLINICAL TRIAL: NCT00258869
Title: Plasma Protein Biomarker Based Diagnostics of Outcome in Sepsis & CAP
Brief Title: Observational Study of Sepsis and Pneumonia to Develop Diagnostic Tests
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Genome Resources (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Duke University (Other); Henry Ford Hospital (Other); Durham VA Medical Center (U.S. Federal Agency); Pfizer (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Stephen F. Kingsmore, President, National Center for Genome Resources
Other Study IDs: 0001; U01AI066569 (NIH)
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2009-01

CONDITIONS: Sepsis; Septicemia; Sepsis Syndrome; Shock, Septic; Community Acquired Pneumonia
Keywords: prospective studies; biological assay; body weights and measures; chemistry, analytical; microchip analytical procedures; spectrum analysis, mass; molecular diagnostic techniques; microbiological techniques; drug administration schedule; data collection; statistics; gene expression profiling; sequence analysis; human experimentation; immunoassay; Trauma severity indices; Glasgow Coma score; Outcome assessment; mortality; computer models; decision modeling; linear models; logistic models; immunologic model; mathematical model; non-linear models; early diagnosis; diagnosis, computer assisted; medical informatics; prognosis; registries; computational biology; systems biology
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome; Shock, Septic; Community-Acquired Pneumonia; Body Weight; Arachnodactyly; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PaxGene whole blood tubes (RNA and DNA), EDTA plasma, serum (subset), microbiologic isolates
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Emergency department patients with sepsis

SUMMARY:
We propose to develop novel diagnostic tests for severe sepsis and community acquired pneumonia (CAP). This program, entitled Community Acquired Pneumonia & Sepsis Outcome Diagnostics (CAPSOD), is a multidisciplinary collaboration involving investigators at six organizations: NCGR; Duke University Medical Center, Durham, NC; Henry Ford Hospital, Detroit, MI; Eli Lilly and Company, Indianapolis, IN; Indiana Centers for Applied Protein Sciences, Indianapolis, IN; and ProSanos Corp., La Jolla, CA.

In the United States, Community Acquired Pneumonia is the sixth leading cause of death and the number one cause of death from infectious diseases. Of the 5.6 million annual cases of CAP, 1.1 million require hospitalization for intensive therapy. Sepsis, commonly known as blood poisoning or bloodstream infection, is the tenth leading cause of death in the US and the number one cause of death in non-cardiac intensive care units. Incidence of sepsis is increasing by 9% each year and mortality rates vary between 25 and 50%. Cost to the US healthcare system exceeds $20 billion each year.

In patients with suspected sepsis or early CAP, rapid identification of patients who will develop severe sepsis or CAP is critical for effective management and positive outcome. The CAPSOD study is designed to identify novel tests for early diagnosis of severe sepsis and CAP. When performed in patients at the earliest stages of disease, these tests will have prognostic value, rapidly identifying those who will have poor outcomes or complicated courses.

CAPSOD will prospectively enroll patients with sepsis and CAP at Duke University Medical Center and Henry Ford Hospital. The study will use advanced bioinformatic, metabolomic, proteomic and mRNA sequencing technologies to identify specific protein changes, or biomarkers, in patient blood samples that predict outcome in sepsis and CAP. Development of biomarker-based tests will permit patient selection for appropriate disposition, such as the intensive care unit, and use of intensive medical therapies, thereby reducing mortality and increasing effectiveness of resource allocation.

DETAILED DESCRIPTION:
3 interdependent aims are proposed to discover and initiate development of novel, in vitro diagnostic tests (IVD) for severe sepsis (SS) and community acquired pneumonia (CAP).

Specific Aim 1: Discovery and initial development of an IVD for early diagnosis of severe sepsis.

In patients with suspected sepsis, early, accurate identification of patients who will develop organ dysfunction (SS) is critical for effective management and positive outcome. While the American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference definitions provide a clinical guide to identifying patients who have SS, we propose to develop a rapid, point-of-care (POC) IVD for early diagnosis of SS. The basis of the proposed IVD will be the measurement of several, host response, plasma proteins. When performed in patients at the earliest stage of sepsis, this test will have prognostic value, rapidly identifying patients who will have poor outcomes or complicated courses.

Availability of this IVD will enable patient selection for appropriate disposition, such as the intensive care unit (ICU), and use of medical therapies, such as early goal-directed therapy (EGDT), thereby reducing mortality and increasing effectiveness of resource allocation. A considerable literature exists of host plasma protein changes during sepsis. Furthermore, in preliminary studies measuring more than 100 host proteins in blood of over 300 patients with SS, we have identified a number of candidate biomarkers of SS. We propose to inventory, replicate and validate the utility of these biomarkers of SS, and to identify novel plasma biomarkers of SS, through literature review and a prospective clinical study employing 2 proteomic technologies (mass spectrometry and multiplexed immunoassays), mass spectrometry-based plasma metabolomics and sequencing of mRNA derived from peripheral blood lymphocytes. We intend to enroll 1200 patients with sepsis (evidence of infection and 2 or more criteria of the systemic inflammatory response syndrome, SIRS) at 3 US tertiary care hospitals and emergency departments (ED), and to monitor their course both by established clinical severity indices (Acute Physiology and Chronic Health Evaluation [APACHE II] and Pneumonia Patient Outcomes Research Team [PORT]scores, and metabolic endpoints such as lactate, base deficit and pH) and ascertainment of complicating events (such as SS, septic shock, acute renal failure (ARF), acute respiratory distress syndrome (ARDS),disseminated intravascular coagulopathy (DIC) and death). It is anticipated that approximately 60% of the patients will develop SS.

Data will be stored in an anonymized, encrypted, web-based patient registry. Bivariable analyses will be performed to identify and validate biomarker differences between groups. Furthermore, we intend to perform predictive modeling using multivariable analyses of the validated biomarkers and derive a biomarker panel and algorithm for early diagnosis of SS. The predictive value of the biomarker panel for early diagnosis of SS will be compared with established prognostic indices, such as metabolic endpoints and APACHE II score. Novel biomarkers of severe CAP will be identified by mass spectrometry of patient EDTA plasma samples. Subject to availability of multiplexed immunoassays, some of these biomarkers will be replicated by immunoassay in the same samples.

During the period of award, a plan for IVD development of the biomarker panel for early diagnosis of SS will be developed. This is anticipated to involve assay optimization and transfer to an existing, validated IVD platform, FDA-regulated IVD development processes, and incorporation of the IVD into an intensive treatment algorithm. The proposed IVD will be an oligoplex assay performed on a single blood sample using immunoassays on an established diagnostic platform with time-to-first result of less than 30 minutes and capable of use in a POC setting, such as an ED or ICU.

Specific Aim 2: Biomarker development for early differentiation of poor outcome in CAP Complications of CAP, including respiratory failure, other organ system failure and severe sepsis, are major determinants of morbidity and mortality. At time of presentation with CAP, accurate identification of patients who will have a complicated course or poor outcome is critical for effective management and positive outcome. In parallel with Specific Aim 1, we propose to identify biomarkers for early diagnosis/prognosis of poor outcome in patients with CAP ("severe CAP"). The biomarkers will be several, host response, plasma proteins that differentiate mild and severe CAP. Early diagnosis of severe CAP will enable patient selection for hospitalization, thereby reducing mortality and increasing effectiveness of resource allocation.

It is anticipated that approximately 33% of the patients enrolled in the Specific Aim 1 clinical study (evidence of infection and two or more SIRS criteria) will have CAP as the underlying infection causing sepsis. Furthermore, it is anticipated that approximately 25% of these CAP patients will develop severe CAP. Specific aim 2 proposes a secondary, separate analysis of all patients enrolled in the Specific Aim 1 clinical study who have CAP in order to identify biomarkers for early diagnosis of severe CAP. We propose to inventory existing candidate biomarkers of severe CAP through literature review. Furthermore, we propose to validate the utility of some of these biomarkers, and to identify a number of novel biomarkers of severe CAP through analysis of the subset of patients in the prospective clinical study who have CAP and employing 2 proteomic technologies (mass spectrometry and multiplexed immunoassays), mass spectrometry-based plasma metabolomics and sequencing of mRNA derived from peripheral blood lymphocytes. Bivariable analyses will be performed to identify plasma biomarker differences between mild and severe CAP. Multivariable analyses will be performed in order to derive a plasma biomarker panel and algorithm for early diagnosis of severe CAP. The biomarker panel for early diagnosis of severe CAP will be compared with established prognostic indices, such as PORT score. Novel biomarkers of severe CAP will be identified by mass spectrometry of patient EDTA plasma samples.

Subject to availability of multiplexed immunoassays, some of these biomarkers will be replicated by immunoassay in the same samples.

During the period of award, a plan for panel validation and IVD development for early diagnosis of severe CAP will be developed. The latter is anticipated to involve assay optimization and transfer to an existing, validated IVD platform, FDA regulated IVD development processes, and incorporation of the IVD into an intensive treatment algorithm. The proposed IVD will be an oligoplex assay performed on a single blood sample using immunoassays on an established diagnostic platform with time-to-first result of less than 30 minutes and capable of use in a POC setting, such as an ED or ICU. This is anticipated to be a product line extension of the SS IVD.

Specific Aim 3: Biomarker development for early differentiation of sepsis and CAP pathogens Currently, initial antimicrobial treatment of sepsis and CAP is empiric. Common etiologic agents in sepsis are gram-positive bacteria (Staphylococcus spp. and Streptococcus spp.), gram-negative bacteria (e.g., Escherichia coli, Klebsiella spp., and Enterobacter spp.), and fungi (Candida spp.). Common etiologic agents in CAP are Streptococcus pneumoniae, Legionella pneumophila, Mycoplasma spp., and viruses. The ability to distinguish these pathogens at time of presentation of sepsis or CAP would potentially allow more targeted rather than broad-spectrum initial therapy. Earlier administration of appropriate antimicrobials would lower patient management cost associated with ineffective therapy and lessen likelihood of antibiotic resistance. We propose to identify host biomarkers for early differentiation of up to 4 common etiologic agents in sepsis and CAP. Our preliminary studies have established proof-of-concept for differentiation between classes of pathogens in sepsis based on specific differences in soluble host proteins in a blood sample. Based on our preliminary studies, it is anticipated that approximately 25% of patients in the Specific Aim 1 clinical study will have a positive blood culture. At least 33 of these patients are anticipated to have S. aureus bacteremia and 20 gram negative bacteremia. Specific Aim 3 proposes to compare plasma samples from patients with S. aureus and gram negative bacteremia in order to identify host biomarkers for early differentiation of specific class agent in sepsis. As in specific aims 1 and 2, bivariable and multivariable analyses of biomarkers is proposed to develop a biomarker panel for early differentiation of staphylococcal and gram-negative sepsis. Similar analysis is proposed to differentiate CAP pathogens. However, given the absence of a high-sensitivity, gold-standard method for determination of causal pathogen in CAP, Specific Aim 3 proposes the more conservative goal of differentiating pneumococcal CAP from atypical CAP based on quantitative differences in host blood biomarkers. The pneumococcal CAP group will be selected from the clinical studydataset based on rigorous criteria: S. pneumoniae from blood or sputum culture or detection of pneumococcal antigen in urine, clinical evidence of CAP and typical (lobar consolidation) chest radiograph. The nonpneumococcal CAP group will be determined by negative pneumococcal cultures and urine antigen, clinical evidence of CAP, and an atypical chest radiograph. It is anticipated that at least 20 patients (15% of the 133 with CAP) will have confirmed pneumococcal CAP and 40 patients (30%) atypical, non-pneumococcal CAP. Biomarkers for differentiation of i. S. aureus bacteremia from gram-negative bacteremia, and ii. pneumococcal CAP from atypical CAP, will be identified by mass spectrometry of patient EDTA plasma samples. Subject to availability of multiplexed immunoassays, some of these biomarkers will be replicated by immunoassay in the same samples. It should be noted that given budget-imposed reduction in patient enrollment of one third from that originally proposed, we are uncertain that sufficient patients will be enrolled for all Specific Aim 3 analyses to be meaningful. We propose to evaluate the group sizes of enrolled patients by specific class agent in order to select two specific comparisons between sepsis and CAP pathogens that are of sufficient size to permit meaningful analysis.

Validation and development of these biomarkers into biomarker panels and rapid, POC, IVD for early differentiation of pathogen in sepsis and CAP is intended, but is beyond the scope of the present proposal. A product line extension of the SS IVD is envisaged. Like the test for early diagnosis of SS, the IVD(s) for early differentiation of CAP and sepsis pathogens will be oligoplex assay(s) performed on single blood sample(s) using immunoassays or other analyte assays.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has known or acute infection or suspected infection AND patient must meet at least 2 of the following 4 criteria to be enrolled

1. A core temperature of >= 38°C (100.4°F) or <= 36°C (96.8°F)
2. Patients > 18 years of age, Heart rate of >= 90 beats/min Patients 13-18 years of age, Heart rate of >= 110 beats/min Patients 6-12 years of age, Heart rate of >= 130 beats/min
3. Patients > 18 years of age, Respiratory rate of >= 20 breaths/min Patients 13-18 years of age, Respiratory rate of >= 14 breaths/min Patients 6-12 years of age, Respiratory rate of >= 18 breaths/min OR PaCO2 of <= 32 mm Hg OR Use of Mechanical Ventilation for an acute respiratory process
4. Patients > 18 years of age, White cell count >= 12,000/mm3 or <= 4,000/mm3 Patients 13-18 years of age, White cell count >= 11,000/mm3 or <= 4,500/mm3 Patients 6-12 years of age, White cell count >= 13,500/mm3 or <= 4,500/mm3 OR A differential count showing > 10% immature neutrophils

Exclusion Criteria:

1. Patient is less than 6 years of age.
2. Patient is not expected to survive 28 days because of uncorrectable medical condition (apart from pneumonia or sepsis), such as poorly controlled neoplasm or other end-stage disease, or patient has active DNR order
3. Human immunodeficiency virus (HIV) infection with a last known CD4 count of <50 mm3
4. Acute presence of a cerebral vascular event, active gastrointestinal hemorrhage, seizure (acute episode), drug overdose, burn injury, trauma
5. Patient is pregnant

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Emergency department patients > 6 years of age
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2005-12; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Death | Day 3
Septic Shock | Day 3
Severe Sepsis | Day 3

SECONDARY OUTCOMES:
Time to death | 28 days
Death | Day 5
Death | Day 7
Death | Day 28
Time to severe sepsis | 28 days
Severe sepsis | Day 5
Severe sepsis | Day 7
Severe sepsis | Day 28
Time to septic shock | 28 days
Septic Shock | Day 5
Septic Shock | Day 7
Septic shock | Day 28
Cryptic shock (ScvO2<65 or Lactate >2.5 and MAP >65 mmHg [>18 years of age] or SBP >90 [<18 years of age]) | Day 3
Time to Cryptic shock (ScvO2<65 or Lactate >2.5 and MAP >65 mmHg [>18 years of age] or SBP >90 [<18 years of age]) | Day 28
Cryptic shock (ScvO2<65 or Lactate >2.5 and MAP >65 mmHg [>18 years of age] or SBP >90 [<18 years of age]) | Day 5
Cryptic shock (ScvO2<65 or Lactate >2.5 and MAP >65 mmHg [>18 years of age] or SBP >90 [<18 years of age]) | Day 7
Cryptic shock (ScvO2<65 or Lactate >2.5 and MAP >65 mmHg [>18 years of age] or SBP >90 [<18 years of age]) | Day 28
Hospitalization | 24 hours
Length of hospital stay | Days
ICU admission | 28 days
Length of ICU admission | Days
Disposition | 28 day
Renal dysfunction | 28 days
Respiratory dysfunction | 28 days
Hematology dysfunction | 28 days
Metabolic dysfunction | 28 days
Renal SOFA score | 28 days
Lung SOFA score | 28 days
Coagulation SOFA score | 28 days
Liver SOFA score | 28 days
CVS SOFA score | 28 dadys
Time to respiratory SOFA Score | 28 days
Time to coagulation SOFA score | 28 days
Time to liver SOFA score | 28 days
Time to CVS SOFA score | 28 days
Time to Renal SOFA score | 28 days
DIC score >5 (modified ISTH scoring system) | 28 days
Time to DIC score > 5 | Days
Development of ALI | 28 days
Development of ARDS | 28 days
Time to ALI | Days
Time to ARDS | Days
Ventilator | 28 days
Ventilator days | Days
MELD score | 28 days
Effect of early goal directed therapy on primary and secondary end-points | 28 days
Effect of Activated Protein C on primary and secondary end-points | 28 days
Effect of stress-dose corticosteroids on primary and secondary end-points | 28 days
Effect of intensive glycemic control on primary and secondary end-points | 28 days
APACHE II score | enrollment
APACHE II score | 24 hours
PRISM III score | enrollment
PRISM III score | 24 hours
SOFA score | enrollment
SOFA score | 24 hours
CAP mortality | Day 3
CAP and severe sepsis | Day 3
CAP and septic shock | Day 3
Severe CAP (ATS criteria) | Day 3
Severe CAP (BTS criteria) | Day 3
Pneumococcal sepsis | Day 7
Staphylococcus aureus sepsis | Day 7
Gram negative rod sepsis | Day 7
Fungal sepsis | Day 7
SeptiFast result | Enrollment
SeptiFast result | 24 hours
Microbiologic culture result | Day 28
Urinary legionella antigen | 7 days
Microbiologic culture | 7 days
CAP, time to death | days
CAP, mortality | Day 5
CAP, mortality | Day 7
CAP, mortality | Day 28
CAP, time to severe sepsis | Days
CAP, severe sepsis | Day 5
CAP, severe sepsis | Day 7
CAP, severe sepsis | Day 28
CAP, time to septic shock | days
CAP, septic shock | Day 5
CAP, septic shock | Day 7
CAP, septic shock | Day 28
Time to severe CAP (ATS and BTS criteria) | Days
Severe CAP (ATS and BTS criteria) | Day 5
Severe CAP (ATS and BTS criteria) | Day 7
Severe CAP (ATS and BTS criteria) | Day 28
CAP, mechanical ventilation | 28 days
CAP, time to mechanical ventilation | Days
CAP, length of mechanical ventilation | Days
CAP, SOFA respiratory score > 2 | 28 days
CAP, respiratory component of severe sepsis criteria | 28 days
CAP, hospitalized | 24 hours
CAP, length of hospitalization | Days
CAP, ICU admission | 28 days
CAP, length of ICU stay | Days
CAP, Disposition | 28 days
CAP, ALI | 28 days
CAP, ARDS | 28 days
CAP, time to ARDS | days
CAP, time to ALI | Days
CAP, PORT score | enrollment
CAP, PORT score | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephen F Kingsmore, MB ChB BAO, Principal Investigator — National Center for Genome Resources; Vance Jr G Fowler, MD, Study Director — Duke University; Emanuel P Rivers, MD, Study Director — Henry Ford Hospital; Christopher W Woods, MD, Study Director — Duke University; Ralph G Corey, MD, Study Director — Duke University; Ronny Otero, MD, Study Director — Henry Ford Hospital; Brian W Grinnell, PhD, Study Director — Eli Lilly and Company; Brian T Edmonds, PhD, Study Director — Eli Lilly and Company; Mu Wang, PhD, Study Director — INCAPS; James R Ludwig, PhD, Study Director — INCAPS
Locations (3):
- United States (3):
  - Henry Ford Hospital, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Durham VA Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Perlee LT, Christiansen J, Dondero R, Grimwade B, Lejnine S, Mullenix M, Shao W, Sorette M, Tchernev VT, Patel DD, Kingsmore SF. Development and standardization of multiplexed antibody microarrays for use in quantitative proteomics. Proteome Sci. 2004 Dec 15;2:9. doi: 10.1186/1477-5956-2-9. eCollection 2004. PMID 15598355
- [Background] Schweitzer B, Roberts S, Grimwade B, Shao W, Wang M, Fu Q, Shu Q, Laroche I, Zhou Z, Tchernev VT, Christiansen J, Velleca M, Kingsmore SF. Multiplexed protein profiling on microarrays by rolling-circle amplification. Nat Biotechnol. 2002 Apr;20(4):359-65. doi: 10.1038/nbt0402-359. PMID 11923841
- [Background] Kingsmore SF, Patel DD. Multiplexed protein profiling on antibody-based microarrays by rolling circle amplification. Curr Opin Biotechnol. 2003 Feb;14(1):74-81. doi: 10.1016/s0958-1669(02)00019-8. PMID 12566005
- [Background] Kaukola T, Satyaraj E, Patel DD, Tchernev VT, Grimwade BG, Kingsmore SF, Koskela P, Tammela O, Vainionpaa L, Pihko H, Aarimaa T, Hallman M. Cerebral palsy is characterized by protein mediators in cord serum. Ann Neurol. 2004 Feb;55(2):186-94. doi: 10.1002/ana.10809. PMID 14755722
- [Background] Kader HA, Tchernev VT, Satyaraj E, Lejnine S, Kotler G, Kingsmore SF, Patel DD. Protein microarray analysis of disease activity in pediatric inflammatory bowel disease demonstrates elevated serum PLGF, IL-7, TGF-beta1, and IL-12p40 levels in Crohn's disease and ulcerative colitis patients in remission versus active disease. Am J Gastroenterol. 2005 Feb;100(2):414-23. doi: 10.1111/j.1572-0241.2005.40819.x. PMID 15667502
- [Background] Heuer JG, Cummins DJ, Edmonds BT. Multiplex proteomic approaches to sepsis research: case studies employing new technologies. Expert Rev Proteomics. 2005 Oct;2(5):669-80. doi: 10.1586/14789450.2.5.669. PMID 16209647
- [Background] Rivers EP, Nguyen HB, Huang DT, Donnino M. Early goal-directed therapy. Crit Care Med. 2004 Jan;32(1):314-5; author reply 315. doi: 10.1097/01.CCM.0000104937.09370.53. No abstract available. PMID 14707615
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Rivers EP, McIntyre L, Morro DC, Rivers KK. Early and innovative interventions for severe sepsis and septic shock: taking advantage of a window of opportunity. CMAJ. 2005 Oct 25;173(9):1054-65. doi: 10.1503/cmaj.050632. PMID 16247103
- [Background] Heuer JG, Sharma GR, Gerlitz B, Zhang T, Bailey DL, Ding C, Berg DT, Perkins D, Stephens EJ, Holmes KC, Grubbs RL, Fynboe KA, Chen YF, Grinnell B, Jakubowski JA. Evaluation of protein C and other biomarkers as predictors of mortality in a rat cecal ligation and puncture model of sepsis. Crit Care Med. 2004 Jul;32(7):1570-8. doi: 10.1097/01.ccm.0000129488.54282.1a. PMID 15241104
- [Background] O'Brien LA, Gupta A, Grinnell BW. Activated protein C and sepsis. Front Biosci. 2006 Jan 1;11:676-98. doi: 10.2741/1827. PMID 16146761
- [Derived] Tsalik EL, Khine A, Talebpour A, Samiei A, Parmar V, Burke TW, Mcclain MT, Ginsburg GS, Woods CW, Henao R, Alavie T. Rapid, Sample-to-Answer Host Gene Expression Test to Diagnose Viral Infection. Open Forum Infect Dis. 2019 Oct 30;6(11):ofz466. doi: 10.1093/ofid/ofz466. eCollection 2019 Nov. PMID 34150923
- [Derived] Tsalik EL, Henao R, Montgomery JL, Nawrocki JW, Aydin M, Lydon EC, Ko ER, Petzold E, Nicholson BP, Cairns CB, Glickman SW, Quackenbush E, Kingsmore SF, Jaehne AK, Rivers EP, Langley RJ, Fowler VG, McClain MT, Crisp RJ, Ginsburg GS, Burke TW, Hemmert AC, Woods CW; Antibacterial Resistance Leadership Group. Discriminating Bacterial and Viral Infection Using a Rapid Host Gene Expression Test. Crit Care Med. 2021 Oct 1;49(10):1651-1663. doi: 10.1097/CCM.0000000000005085. PMID 33938716
- [Derived] Tsalik EL, Langley RJ, Dinwiddie DL, Miller NA, Yoo B, van Velkinburgh JC, Smith LD, Thiffault I, Jaehne AK, Valente AM, Henao R, Yuan X, Glickman SW, Rice BJ, McClain MT, Carin L, Corey GR, Ginsburg GS, Cairns CB, Otero RM, Fowler VG Jr, Rivers EP, Woods CW, Kingsmore SF. An integrated transcriptome and expressed variant analysis of sepsis survival and death. Genome Med. 2014 Nov 26;6(11):111. doi: 10.1186/s13073-014-0111-5. eCollection 2014. PMID 25538794
- [Derived] Glickman SW, Cairns CB, Otero RM, Woods CW, Tsalik EL, Langley RJ, van Velkinburgh JC, Park LP, Glickman LT, Fowler VG Jr, Kingsmore SF, Rivers EP. Disease progression in hemodynamically stable patients presenting to the emergency department with sepsis. Acad Emerg Med. 2010 Apr;17(4):383-90. doi: 10.1111/j.1553-2712.2010.00664.x. PMID 20370777
- [Derived] Tsalik EL, Jones D, Nicholson B, Waring L, Liesenfeld O, Park LP, Glickman SW, Caram LB, Langley RJ, van Velkinburgh JC, Cairns CB, Rivers EP, Otero RM, Kingsmore SF, Lalani T, Fowler VG, Woods CW. Multiplex PCR to diagnose bloodstream infections in patients admitted from the emergency department with sepsis. J Clin Microbiol. 2010 Jan;48(1):26-33. doi: 10.1128/JCM.01447-09. Epub 2009 Oct 21. PMID 19846634